CLINICAL TRIAL: NCT06732037
Title: Effect of Kinetic Control Training on Flexion Relaxation Phenomenon and Craniovertebral Angle in Cervical Radiculopathy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Adel Ibrahim Farahat, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004384
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy program (Active Comparator): It consists of thirty patients with cervical radiculopathy. They will receive conventional physical therapy program.
  Interventions: Other: Conventional physical therapy program
- Conventional physical therapy program + Kinetic control training (Experimental): It consists of thirty patients with cervical radiculopathy. They will receive conventional physical therapy program plus kinetic control training.
  Interventions: Other: Conventional physical therapy program; Other: Kinetic control training

INTERVENTIONS:
Other: Conventional physical therapy program — The conventional physical therapy program will be received for 8 weeks by the two groups. It includes the application of moist heat using a hot pack for ten minutes, followed by continuous ultrasound therapy operated at a frequency of 1 MHz and an intensity of 1.5 W/cm² for five minutes. Transcutaneous Electrical Nerve Stimulation (TENS) will also be utilized, with its development and application based on the Gate Control Theory. TENS will be applied for twenty minutes, with electrodes positioned on either side of the neck at the level of pain, using a pulse rate ranging from 2 to 50 Hz.
Other: Kinetic control training — The Kinetic Control Retraining Program will be received for 8 weeks by the experimental group. It focuses on addressing uncontrolled movement (UCM) and muscle synergy retraining. UCM retraining starts with patient education on movement deficiencies, their symptoms, and adherence to training. Movement coordination is retrained in test positions, progressing to challenging ones using feedback from mirrors, walls, or hands. Corrections focus on lower cervical flexion, upper cervical extension, mid-cervical translation/extension, side-bending, and rotation, emphasizing controlled dissociation in supported and unsupported postures. Muscle synergy retraining targets global stabilizers (e.g., deep neck flexors and extensors) and mobilizers (e.g., sternocleidomastoid and suboccipital muscles) to enhance coordination, stability, and motor control.
  Arms: Conventional physical therapy program + Kinetic control training

SUMMARY:
The purpose of the study is to determine the effect of kinetic control training on flexion relaxation phenomenon and craniovertebral angle in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
Neck pain is a major health issue with high rates of recurrence. The current literature suggests people with cervical pain have altered movement control strategies and that these changes are associated with pain and disability.

These altered strategies will influence the control of movement which can present as both uncontrolled translatatory movement and uncontrolled range or physiological motion. Either movement dysfunction will present clinically as areas of relative flexibility (increase in translational movement) or areas of relative stiffness.

Changes in alignment in the cervical spine may result in a forward head posture position demonstrating an increase in low cervical flexion.

The greater the forward head posture, the greater the disability. Regions and segments of less mobility have been noted in the cervical spine which will present clinically as regions of relative stiffness.

Disturbance in neck flexor synergy has been commonly observed in patients with neck pain. This disturbed neck flexor synergy presents as altered pattern of muscle activity, where impairment in deep cervical flexors appears to be compensated by increased activity in superficial muscles (sternocleidomastoid and anterior scalene) and it is also reported that the amplitude of upper trapezius and cervical extensors have been dramatically increased among those patients. Such impairments may contribute to the development of pain and disability in patients with neck pain.

The Kinetic Control retraining strategy consists of patient education about his uncontrolled movement, retraining the coordination of movement direction control and muscle synergy retraining. Movement retraining interventions that are matched to correcting specific impairments can restore movement and performance solutions, elevating movement health and the quality of life it supports.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be referred from neurologist with the diagnosis cervical spondylosis.
2. Patients will be included if they have unilateral radiculopathy due to spondylotic changes of the lower cervical spine (C5-C6 and C6-C7).
3. Duration of symptoms is more than three months to avoid acute stage of inflammation.
4. Patient's age ranged from 40 to 55 years.
5. Patients from both sexes.
6. Body mass index of all patients is ranged from 25-30 kg/m2.
7. Patients will be screened prior to inclusion by measuring the craniovertebral angle, if the angle was less than 50, then a participant will be referred to the study

Exclusion Criteria:

1. Spinal canal stenosis.
2. Rheumatoid arthritis.
3. Vertebrobasilar insufficiency.
4. Spinal instability due to structural cause e.g., spondylolisthesis.
5. Systemic disease (cardiovascular, infectious and/or metabolic disease that could interrupt exercises).
6. Spinal tumors.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-22 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain | 8 weeks
  The Visual analogue scale is used for pain assessment. In this scale, pain is rated from 0 to 100 mm, in which the 0 represented no pain and100 Represented maximum pain tolerance. Subjects are indicated the best number described their pain.
Assessment of craniovertebral angle (CVA) | 8 weeks
  Markus Bader ruler (MB ruler) is a computer-based objective tool that measure angles and distances. Reflective markers will be placed on participants' anatomical landmarks and a photograph will be taken. The photograph will be uploaded to a computer and the MB ruler software will be used to calculate the CVA.
Assessment of flexion relaxation phenomenon using surface electromyography | 8 weeks
  Cervical flexion relaxation phenomenon (FRP) is a myoelectric silence of neck extensor muscles which occurs after a certain degree of flexion. Patients will accomplish cervical flexion and extension from a neutral position in four phases in the sitting position. The surface electromyography activity of cervical erector spinae (CES) will be recorded in each phase.

SECONDARY OUTCOMES:
Assessment of disability | 8 weeks
  The Neck Disability Index (NDI), a modification of the Oswestry Low Back Pain Disability Index, is a widely used instrument for measuring self-rated disability due to neck pain, utilized by clinicians and researchers alike. It is a condition-specific, patient-completed functional status questionnaire consisting of 10 items: pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored from 0 to 5, with a maximum score of 50. The total score can be multiplied by two to yield a percentage score, providing a standardized measure of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Samir Mohamed Fayez, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt